CLINICAL TRIAL: NCT05552443
Title: Identification of the Optimal Analgesic Dose of Intrathecal Hydromorphone for Pediatric Patients Undergoing Posterior Spine Surgery for Idiopathic Scoliosis
Brief Title: A Study of Intrathecal Hydromorphone for Pediatric Idiopathic Scoliosis Repair
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study participant #27 had a related adverse event that prompted interim data analysis and additional study participants were not sought.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kathryn (Katie) S. Handlogten, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 22-006823
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Pain Control
Keywords: Posterior Spine Surgery; Pediatric Idiopathic Scoliosis Repair
MeSH Terms: conditions — Agnosia | interventions — Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Intrathecal Hydromorphone 2.5 mcg/kg (Experimental): Subjects undergoing posterior spinal surgery will receive 2.5 mcg/kg hydromorphone in the intrathecal space at the low lumbar level
  Interventions: Drug: Hydromorphone 2.5 mcg/kg
- Intrathecal Hydromorphone 2.75 mcg/kg (Experimental): Subjects undergoing posterior spinal surgery will receive 2.75 mcg/kg hydromorphone in the intrathecal space at the low lumbar level
  Interventions: Drug: Hydromorphone 2.75 mcg/kg
- Intrathecal Hydromorphone 3 mcg/kg (Experimental): Subjects undergoing posterior spinal surgery will receive 3 mcg/kg hydromorphone in the intrathecal space at the low lumbar level
  Interventions: Drug: Hydromorphone 3 mcg/kg
- Intrathecal Hydromorphone 3.25 mcg/kg (Experimental): Subjects undergoing posterior spinal surgery will receive 3.25 mcg/kg hydromorphone in the intrathecal space at the low lumbar level
  Interventions: Drug: Hydromorphone 3.25 mcg/kg
- Intrathecal Hydromorphone 3.5 mcg/kg (Experimental): Subjects undergoing posterior spinal surgery will receive 3.5 mcg/kg hydromorphone in the intrathecal space at the low lumbar level
  Interventions: Drug: Hydromorphone 3.5 mcg/kg
- Intrathecal Hydromorphone 4 mcg/kg (Experimental): Subjects undergoing posterior spinal surgery will receive 4 mcg/kg hydromorphone in the intrathecal space at the low lumbar level
  Interventions: Drug: Hydromorphone 4 mcg/kg
- Intrathecal Hydromorphone 4.5 mcg/kg (Experimental): Subjects undergoing posterior spinal surgery will receive 4.5 mcg/kg hydromorphone in the intrathecal space at the low lumbar level
  Interventions: Drug: Hydromorphone 4.5 mcg/kg
- Intrathecal Hydromorphone 5 mcg/kg (Experimental): Subjects undergoing posterior spinal surgery will receive 5 mcg/kg hydromorphone in the intrathecal space at the low lumbar level
  Interventions: Drug: Hydromorphone 5 mcg/kg

INTERVENTIONS:
Drug: Hydromorphone 2.5 mcg/kg — 2.5 mcg/kg intrathecal
  Arms: Intrathecal Hydromorphone 2.5 mcg/kg
Drug: Hydromorphone 2.75 mcg/kg — 2.75 mcg/kg intrathecal
  Arms: Intrathecal Hydromorphone 2.75 mcg/kg
Drug: Hydromorphone 3 mcg/kg — 3 mcg/kg intrathecal
  Arms: Intrathecal Hydromorphone 3 mcg/kg
Drug: Hydromorphone 3.25 mcg/kg — 3.25 mcg/kg intrathecal
  Arms: Intrathecal Hydromorphone 3.25 mcg/kg
Drug: Hydromorphone 3.5 mcg/kg — 3.5 mcg/kg intrathecal
  Arms: Intrathecal Hydromorphone 3.5 mcg/kg
Drug: Hydromorphone 4 mcg/kg — 4 mcg/kg intrathecal
  Arms: Intrathecal Hydromorphone 4 mcg/kg
Drug: Hydromorphone 4.5 mcg/kg — 4.5 mcg/kg intrathecal
  Arms: Intrathecal Hydromorphone 4.5 mcg/kg
Drug: Hydromorphone 5 mcg/kg — 5 mcg/kg intrathecal
  Arms: Intrathecal Hydromorphone 5 mcg/kg

SUMMARY:
The purpose of this study is to identify a dose of intrathecal hydromorphone (opioid pain medicine) that optimizes pain control but minimizes side effects historically seen with this class of pain medications.

DETAILED DESCRIPTION:
This study is a sequential coin based up-down dose allocation method with the goal of identifying the ED90 for intrathecal hydromorphone (ITH) in idiopathic adolescent scoliosis repair via the posterior approach. A starting dose of 3.5 mcg/kg of hydromorphone was determined by current practice at the institution as well as upon review of available literature of previously used ITM doses in pediatric spine patients. Subsequent participants will receive higher (step "up") or lower (step "down") from this starting dose. Steps "down" from the starting dose will be smaller than steps "up" to ensure maintenance of adequate analgesia and to allow more accurate estimate of the optimal dose should it decrease beyond our starting dose. Steps "up" from the starting dose were chosen based on commonly used weight-based doses in our current practice. A maximum dose of 400 mcg, despite patient weight, was determined based on expert consensus and review preparatory to research query. The anesthesiologist covering the case (high lumbar or thoracic corrections) or the surgeon (low lumbar corrections) will administer the medication at the low lumbar level.

ITH dose adjustments for subsequent study patients will be based on the efficacy of the dose used with the prior patient. Efficacious ITH administration will be defined as all NRS scores ≤5 within the first 18 hours after administration (binary outcome). If the NRS score was >5 within 18 hours or if the patient required supplemental opioid administration for pain control (suggestive of insufficient analgesia), the dose will be increased for the next enrolled study patient. If the pain score remains ≤5 within 18 hours of opioid administration, the next patient will receive the next lower dose or the same dose as the previous patient. Patients excluded after randomization will be removed from the study.

ELIGIBILITY:
Inclusion Criteria:

- Undergoing spinal surgery with a posterior approach for idiopathic scoliosis.

Exclusion criteria:

* Patients with pre-surgical elevated pain scores (≥ 3/10 on Numeric Rating Scale (NRS)), history of chronic pain, or pre-surgical opioid use will not be included.
* Patients with contraindications to spinal anesthesia (anatomical abnormality or elevated bleeding or infection risks) will not be included.
* Patients for whom the protocol is violated (inability to perform postoperative data collection), or the study/procedure was aborted will not be included in analysis.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-10-27 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 18 hours after intrathecal hydromorphone administration
  Reported by the patient using an 11-point numeric visual analogue scale (NRS) with 0=no pain and 10=worst pain ever

SECONDARY OUTCOMES:
Incidence of need for dual anti-pruritic agents | 24 postoperative hours
  Number of subjects needing dual anti-pruritic agents (Nubain or naloxone (beyond the protocol infusion rate of 0.25 mcg/kg/min))
Maximum pain scores | 24 hours after intrathecal hydromorphone administration
  Highest pain score reported during the first 24 hours after intrathecal opioid administration. Reported by the patient using an 11-point numeric visual analogue scale (NRS) with 0=no pain and 10=worst pain ever.
OME consumption | 24 hours after intrathecal hydromorphone administration
  Total oral morphine equivalents (OME) consumption
Incidence of antiemetic use postoperatively | 24 postoperative hours
  Number of subjects to require antiemetic medications used to prevent or treat nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Handlogten, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials